CLINICAL TRIAL: NCT02768051
Title: EP Dynamics (EPD) Research First In Man Clinical Study
Brief Title: Evaluation of the Safety, Feasibility and Usability of the EPD D700 System in Atrial Flutter Ablation Procedures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision of the management
Sponsor: EPD Solutions, A Philips Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN-D700-001
Record Dates: First submitted 2016-05-01; First posted 2016-05-11 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Atrial Flutter
MeSH Terms: conditions — Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AF Ablation Intervention (Experimental): Subjects who are scheduled to undergo ablation procedure due to atrial flutter.
  Interventions: Procedure: AF Ablation

INTERVENTIONS:
Procedure: AF Ablation

SUMMARY:
Demonstrate the safety, feasibility and usability of the EPD D700 system, for the first time in humans, in subjects undergoing ablation for the treatment of atrial flutter.

Prospective, single-center, non-randomized, open label, single arm study. Ten consented subjects who are scheduled to undergo ablation due to atrial flutter. All subjects will undergo baseline assessment; intervention (standard fluoroscopy guided RF ablation procedure) and post procedure follow up. All subjects will have a follow up visit within 24 hours post procedure.

DETAILED DESCRIPTION:
All procedures will be performed under standard fluoroscopic guidance for the treatment of atrial flutter ablation procedure, and the D700 system will be used additionally to demonstrate system safety, feasibility and usability.

The entire procedure will be conducted as customary, using standard and approved off- the-shelf equipment (body surface electrodes, diagnostic and irrigated ablation catheters, RF generator and recording system), in a completely clinically independent manner from the D700 system that will merely be a 'silent witness'. The operator will neither use nor rely on any of the D700 system output for clinical decision making.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age.
2. Subject or authorized representative, signed a written Informed Consent form to participate in the study, prior to any study related procedures.
3. Subject is willing to comply with the protocol requirements and return to the treatment center for all required clinical evaluations.
4. Subject is generally in good health.
5. A female subject is eligible if not of child bearing potential or has a negative pregnancy test within the previous 7 days.
6. Subject is deemed amenable to therapeutic ablation for atrial flutter.

Exclusion Criteria:

1. Any planned surgical or endovascular intervention within 30 days before or after the index procedure.
2. Subject is enrolled in another drug or device study protocol that has not reached its primary endpoint.
3. Patient had experienced previous stroke (TIA or CVA).
4. Patient has a pacemaker.
5. Thrombi detected in the heart.
6. Known marked valvar insufficiency.
7. Life expectancy less than 12 months.
8. Known severe renal insufficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05 (Estimated); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Safety Endpoint - Any intra-procedural or immediate post-procedure complications. | Intra-procedural or immediate post-procedure

SECONDARY OUTCOMES:
Feasibility - Freedom from any impact on current workflow or clinical efficacy. | Intra-procedural or immediate post-procedure
Usability - Correct visualization of the catheter spatial location (map reference). | Intra-procedural or immediate post-procedure

IPD SHARING:
Plan to Share IPD: Undecided